CLINICAL TRIAL: NCT01907503
Title: Adaptation of Locomotor Activity in Patients Suffering From Hip OA - Analysis of This Adaptation as a Prognostic Criterion for Future Disease Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Maillefert PHRC R 2004
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Primary Hip Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with Primary hip osteoarthritis (Other): Patients with Primary hip osteoarthritis
  Interventions: Procedure: Evaluation of the balance of force platform
- Healthy volunteer (Other): Healthy volunteer
  Interventions: Procedure: Evaluation of the balance of force platform

INTERVENTIONS:
Procedure: Evaluation of the balance of force platform

SUMMARY:
To assess the prognostic value of a characteristic evaluation of gait in persons suffering from hip OA for subsequent indications for THR.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 45 and 75 years Suffering from primary hip osteoarthritis defined according to ACR criteria who presented pain in the hip for at least one month in the preceding 3 months Radiological stage II, III or IV hip OA according to the Kellgren and Lawrence classification Patients able to understand simple instructions des packaging instructions, to give their written informed consent.

Exclusion Criteria:

* Indication for THR at the time of inclusion. Pregnant or breast-feeding women Alzheimer's disease Chronic respiratory insufficiency with clinical manifestations Parkinson's disease Motor neuron disease Major musculo-skeletal disorder (other than hip OA) Severe non-stabilised diabetes Non-stabilised hypertension Hip OA inflammation flare Rapidly-destructive hip OA Radiography to evaluate structural evolution of the disease done more than 12 months previously Presence of OA in another joint, or another osteoarticular or periarticular disease of the lower limbs with, in the opinion of the patient, disability due to this other disease that is greater than the disability caused by the hip OA.

Spine disease causing gait disturbance (radiculalgia, lumbar canal stenosis,… with, in the opinion of the patient, disability due to this other disease that is greater than the disability caused by the hip OA.)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-02; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
locomotor activity | participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Derived] Yang Q, Ji X, Zhang Y, Du S, Ji B, Zeng W. An interpretable machine learning approach for predicting and grading hip osteoarthritis using gait analysis. BMC Musculoskelet Disord. 2025 Jul 1;26(1):580. doi: 10.1186/s12891-025-08911-6. PMID 40597862
- [Derived] Moissenet F, Naaim A, Ornetti P, Bourredjem A, Binquet C, Morisset C, Gouteron A, Maillefert JF, Laroche D. Is the Pelvis-Thorax Coordination a Valuable Outcome Instrument to Assess Patients With Hip Osteoarthritis? Front Bioeng Biotechnol. 2020 Jan 23;7:457. doi: 10.3389/fbioe.2019.00457. eCollection 2019. PMID 32039174